CLINICAL TRIAL: NCT05676502
Title: Nasal High Flow (NHF) in COPD - Effects on Ventilation With Asymmetrical Nasal Cannulas (NHFDuet)
Brief Title: Effects on Ventilation With NHF and Asymmetrical Nasal Cannulas
Acronym: NHFDuet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kliniken Essen-Mitte (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Principal Investigator, Georg Nilius, Prof. Dr. med, Head of Department of Pneumology, PI, Kliniken Essen-Mitte
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NHFDuet 2022
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Nasal High Flow (NHF); High Flow Nasal Cannula (HFNC); Optiflow; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal High Flow with Optiflow M cannula (Active Comparator): Nasal high flow treatment 35L/min with the standard symmetric nasal cannula (Optiflow M)
  Interventions: Device: AIRVO 2
- Nasal High Flow with Optiflow Duet Cannula (Active Comparator): Nasal high flow treatment 35L/min with the asymmetric nasal cannula (Optiflow Duet)
  Interventions: Device: AIRVO 2

INTERVENTIONS:
Device: AIRVO 2 — Patients with chronic obstructive pulmonary disease and chronic respiratory failure use Nasal High Flow therapy during daytime sessions of 1.5 h.
  Other Names: Nasal High Flow

SUMMARY:
The aim of this controlled randomized crossover study is to compare the physiological effects of nasal high flow therapy (NHF) with 2 different nasal cannulas in patients with exacerbated chronic obstructive pulmonary disease (ECOPD) and chronic respiratory failure.

20 patients will be treated with NHF therapy (Airvo, Fisher&Paykel Healthcare, NZ) during wakefulness. Physiological measuremends will take place over three perdiods (visits). One period without NHF, one with NHF via standard cannula (Optiflow M) and one with asymmetrical cannula (Optiflow Duet) in randomised order.

DETAILED DESCRIPTION:
Background: Nasal High Flow (NHF) therapy had shown to increase airway pressure, reduce dead space, and improve mucociliary clearance and gas exchange in patients suffering from chronic obstructive pulmonary disease (COPD). The long-term and short-term physiological aspects of NHF are subject of ongoing research. Different flow rates and cannula sizes have been studied and found to yield different therapeutic effects. Larger sized cannulas tend to seal the nares and produce increased positive airway pressure, while smaller cannulas increase the washout effect. Currently, a new cannula is available, with one smaller and one larger opening (Optiflow+ Duet, Fisher&Paykel Healthcare, NZ).

Procedure: Following a baseline period without high flow therapy, NHF (35L/min) will be applied via the nasal cannula (Duet or Standard in randomized order). After a wash out phase, the NHF interface will be replaced for another measurement with the respective other cannula (Standard or Duet).

Respiratory rate, tidal volume, minute ventilation, inhalation to exhalation ratio (Ti/Te), transcutaneous pCO2 and intercostal EMG will be recorded during each partial measurement.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with COPD GOLD 3 and 4 in stable phase after acute exacerbation
* Inpatients with COPD GOLD (2, 3 and 4)
* Informed Consent

Exclusion Criteria:

* Acute respiratory insuffiency with respiratory acidosis (pH<7.35)
* Severe acute physical disease, that do not allow the subject to participate in a clinical trial
* Language, cognitive, or other barriers that make study participation impossible
* Pregnancy or Nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in minute ventilation (MV) comparing arm 1 and 2 | 1.5 hours
  Respiratory effort measured with calibrated RIP system (Respitrace QDC; Viasys Services, Lakeland, FL), MV is calculated. Unit is L

SECONDARY OUTCOMES:
Change in respiratory rate (RR) comparing arm 1 and 2 | 1.5 hours
  Respiratory effort measured with calibrated RIP system (Respitrace QDC; Viasys Services, Lakeland, FL), RR is calculated. Unit is breath per minute
Change in inhalation to exhalation ratio (Ti/Te) comparing arm 1 and 2 | 1.5 hours
  Respiratory effort is measured with calibrated RIP system (Respitrace QDC; Viasys Services, Lakeland, FL), (Ti/Te) is calculated.

OTHER OUTCOMES:
Change oin intercostal surface EMG (surfEMG) comparing arm 1 and 2 | 1.5 hours
  SurfEMG is measured with EMG system (ADInstruments, NZ), it represents the neural respiratory drive, max ampltude of EMG, unit is mV

CONTACTS AND LOCATIONS:
Locations (1):
- Georg N Nilius, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No